CLINICAL TRIAL: NCT04091438
Title: A Phase 1b Randomized, Double-Blind, Placebo-Controlled, Crossover Study of a Single Intravenous Infusion Dose of TAK-925 in Patients With Idiopathic Hypersomnia
Brief Title: A Study of a Single Intravenous Infusion Dose of TAK-925 in Participants With Idiopathic Hypersomnia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-925-2002; U1111-1238-3314 (Registry Identifier: WHO); JapicCTI-195087 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Results first posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2022-11

CONDITIONS: Idiopathic Hypersomnia
Keywords: Drug therapy
MeSH Terms: conditions — Idiopathic Hypersomnia | interventions — TAK-925

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAK-925 Dose A + Placebo (Experimental): TAK-925 112 milligram (mg), 9-hour intravenous infusion once on Day 1, Treatment Period 1 followed by 24 hours wash-out period, followed by TAK-925 placebo-matching 9-hour intravenous infusion once on Day 3, Treatment Period 2.
  Interventions: Drug: TAK-925; Drug: TAK-925 Placebo
- Placebo + TAK-925 Dose A (Placebo Comparator): TAK-925 placebo-matching 9-hour intravenous infusion once on Day 1, Treatment Period 1 followed by 24 hours wash-out period, followed by, TAK-925 112 mg, 9-hour intravenous infusion once on Day 3, Treatment Period 2.
  Interventions: Drug: TAK-925; Drug: TAK-925 Placebo

INTERVENTIONS:
Drug: TAK-925 — TAK-925 IV infusion.
Drug: TAK-925 Placebo — TAK-925 placebo-matching IV infusion.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of administering a single intravenous (IV) infusion dose of TAK-925 to adult participants with idiopathic hypersomnia (IH).

DETAILED DESCRIPTION:
The drug being tested in this study in participants with IH is called TAK-925. The study will have 2-treatment crossover groups. The study will evaluate the pharmacokinetics (PK), pharmacodynamics (PD), safety, and tolerability of a single intravenous (IV) dose of Dose A in participants with IH.

The study will enroll 40 patients. Participants will be randomly assigned to one of the two treatment sequence groups as indicated below:

* TAK-925 + Placebo
* Placebo + TAK-925

On Day 1 of each treatment period, TAK-925 or placebo will be administered as a single 9-hour IV infusion.

The multicenter study will be conducted in the United States and Japan. The overall duration of treatment in this study is approximately 41 days including screening up to 28 days, confinement for 6 days and end of study follow up telephone call on Study Day 11.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of IH, as defined by the International Classification of Sleep Disorders-3 (ICSD-3) as verified by a previous nocturnal polysomnography (nPSG) and multiple sleep latency test (MSLT) study performed within the last 10 years.
2. Onset of hypersomnia between 10 and 30 years of age.
3. Seven consecutive days of actigraphy supported by a sleep diary obtained prior to the nPSG (Study Day -2) shows an average nightly sleep duration of greater than or equal to (>=) 420 minutes during the participant's normal nocturnal sleep period.
4. nPSG (Study Day -2) demonstrates that participant does not have other comorbid sleep disorders or clinically significant nocturnal hypoxemia (oxygen saturation ≤80% for ≥5% of total sleep time) and that their Apnea-Hypopnea Index (AHI) is less than or equal to (<=) 10 per hour, their periodic limb movement arousal index (PLMAI) <=15/hour, and that their total sleep time is >=6.5 hours.
5. Participants taking medication for treatment of excessive daytime sleepiness (EDS) must be willing to discontinue medication prior to randomization into the study.
6. Body mass index (BMI) of 18 through 33 kilogram per square meter (kg/m^2) inclusive.
7. Epworth Sleepiness Scale (ESS) score >=11 at screening and on Day -2.
8. Blood pressure (BP) must be <140 mmHg (systolic) and <90 mmHg (diastolic) at screening and Study Day -2.

Exclusion Criteria:

1. Average nightly sleep duration is <=8 hours (480 minutes) and has insufficient sleep syndrome as evidenced by sleeping >2 hours/night more on "off-days" relative to "work days" as determined by actigraphy and sleep diary obtained prior to the nPSG (Study Day -2).
2. Positive urine screen for drugs of abuse and/or positive alcohol test at screening and Study Day -2.
3. Resting heart rate (HR) outside of the range of 40 to 90 beats pper minute (bpm) off stimulants.
4. Screening electrocardiogram (ECG) reveals a QT interval with Fridericia correction method >450 ms (men) or >470 ms (women).
5. Usual bedtime later than 24:00 (midnight) or an occupation requiring nighttime shift work or variable shift work within the past 6 months, or travel with significant jet lag within 14 days before Study Day -2.
6. History of a sleep disorder other than IH, based on interviews at the screening visit, such as obstructive sleep apnea (OSA), restless legs syndrome, or periodic limb movements of sleep (PLMS) associated with arousals.
7. Use of any over-the-counter (OTC) or prescription medications with stimulating properties within 7 days prior to dosing or 5 half-lives (whichever is longer) that could affect the evaluation of EDS or use of sodium oxybate within 3 months of screening.
8. Nicotine dependence that is likely to have an effect on sleep (e.g., a participant who routinely awakens at night to smoke) and/or an unwillingness to discontinue all smoking and nicotine use during the confinement portion of the study (Day -2 to Day 4).
9. Caffeine consumption of more than 600 mg/day for 7 days before Study Day 1 (1 serving of coffee is approximately equivalent to 120 mg of caffeine) and/or unwilling to discontinue all caffeine during the confinement portion of the study (Day -2 to Day 4).
10. Alcohol use that is likely to have an effect on sleep and/or an unwillingness to discontinue all alcohol use from 72 hours before check-in through discharge on Study Day 4.
11. History of epilepsy or seizures, including having had a single seizure or a history of childhood febrile seizures or has a clinically significant history of head trauma.
12. Answered "YES" on Questions 4 or 5 on the Suicidal Ideation subscale of the Columbia Suicide Severity Rating Scale (C-SSRS) at screening (defined period as 3 months prior to screening) or evidence of suicidal behavior within 6 months of screening as measured by the Suicidal Behavior subscale of the C-SSRS.
13. Diagnosis of major depressive disorder (DSM-5), within the past 6 months or Beck Depression Inventory II (BDI-II) total score of >16 at the screening visit.
14. History of cerebral ischemia, transient ischemic attack, intracranial aneurysm, or arteriovenous malformation.
15. Known coronary artery disease, a history of myocardial infarction, angina, cardiac rhythm abnormality, or heart failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-01-26 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (22):
- United States (20):
  - Wright Clinical Research, Alabaster, Alabama
  - Pulmonary Associates Clinical Trials, Glendale, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Stanford School of Medicine, Redwood City, California
  - Pacific Research Network, Inc, San Diego, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Delta Waves Sleep Disorders and Research Center, Colorado Springs, Colorado
  - St Francis Medical Institute, Clearwater, Florida
  - MD Clinical, Hallandale, Florida
  - Research Centers of America, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Pulmonary Disease Specialists, PA, d/b/a PDS Research, Kissimmee, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Global Research Associates, Stockbridge, Georgia
  - Helene A. Emsellem, MD PC trading as "The Center for Sleep & Wake Disorders", Chevy Chase, Maryland
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Sleep Therapy & Research Center, San Antonio, Texas
- Japan (2):
  - SOUSEIKAI PS Clinic, Hakata-ku, Fukuoka
  - Sumida Hospital, Sumida-ku, Tokyo-To

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Mignot E, Bogan RK, Emsellem H, Foldvary-Schaefer N, Naylor M, Neuwirth R, Faessel H, Swick T, Olsson T. Safety and pharmacodynamics of a single infusion of danavorexton in adults with idiopathic hypersomnia. Sleep. 2023 Sep 8;46(9):zsad049. doi: 10.1093/sleep/zsad049. PMID 36883238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 13 investigative sites in the United States and Japan from 26 January 2020 to 23 November 2020.
Pre-assignment Details: Participants with idiopathic hypersomnia (IH) were enrolled in one of the two treatment sequences of this 2-period crossover study to receive TAK-925 112 milligram (mg) infusion or placebo.
Groups:
- Sequence 1: TAK 925 112 mg + Placebo: TAK-925 112 mg, infusion, intravenously, once on Day 1 (Study Day 1) of Treatment Period 1, followed by 24 hours washout period, further followed by placebo, infusion, intravenously, once on Day 1 (Study Day 3) of Treatment Period 2.
- Sequence 2: Placebo + TAK-925 112 mg: Placebo, infusion, intravenously, once on Day 1 (Study Day 1) of Treatment Period 1, followed by 24 hours washout period, further followed by TAK-925 112 mg, intravenously, once on Day 1 (Study Day 3) of Treatment Period 2.
Period: Treatment Period 1 (1 Day)
Arm/Group | Sequence 1: TAK 925 112 mg + Placebo | Sequence 2: Placebo + TAK-925 112 mg
Started | 14 | 14
Treated | 13 | 14
Completed | 13 | 14
Not Completed | 1 | 0
Not completed — Other | 1 | 0
Period: Washout Period (1 Day)
Arm/Group | Sequence 1: TAK 925 112 mg + Placebo | Sequence 2: Placebo + TAK-925 112 mg
Started | 13 | 14
Completed | 13 | 12
Not Completed | 0 | 2
Not completed — Protocol deviation | 0 | 1
Not completed — Other | 0 | 1
Period: Treatment Period 2 (1 Day)
Arm/Group | Sequence 1: TAK 925 112 mg + Placebo | Sequence 2: Placebo + TAK-925 112 mg
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: TAK 925 112 mg + Placebo | Sequence 2: Placebo + TAK-925 112 mg | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (9.97) | 31.5 (7.91) | 31.7 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 11 | 14 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 3 | 1 | 4
  United States of America | 10 | 13 | 23
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 165.18 (8.077) | 170.10 (9.924) | 167.73 (9.253)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 64.33 (11.501) | 78.88 (16.067) | 71.87 (15.652)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 23.47 (3.336) | 27.02 (3.597) | 25.31 (3.857)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least One Treatment-emergent Adverse Event (TEAE)
Time Frame: Study Day 1 up to Study Day 11
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo, infusion, intravenously, once on Day 1 (Study Day 1 or Study Day 3) of Treatment Period 1 or 2.
- TAK-925 112 mg: TAK-925 112 mg, infusion, intravenously, once on Day 1 (Study Day 1 or Study Day 3) of Treatment Period 1 or 2.
Arm/Group | Placebo | TAK-925 112 mg
Number analyzed (Participants) | 27 | 25
percentage of participants | 14.8 | 40.0

2. Primary Outcome: Percentage of Participants With Markedly Abnormal Criteria for Clinical Safety Laboratory Tests
Time Frame: Study Day 1 up to Study Day 11
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Groups:
- TAK 925 112 mg: TAK-925 112 mg, infusion, intravenously, once on Day 1 (Study Day 1 or Study Day 3) of Treatment Period 1 or 2.
Arm/Group | Placebo | TAK 925 112 mg
Number analyzed (Participants) | 27 | 25
percentage of participants | 3.7 | 0

3. Primary Outcome: Percentage of Participants With Markedly Abnormal Criteria for Vital Sign Measurements
Time Frame: From Predose up to Study Day 4
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-925 112 mg
Number analyzed (Participants) | 27 | 25
percentage of participants
  Systolic Blood Pressure: less than (<) 90 millimeter of mercury (mmHg) | 14.8 | 12.0
  Systolic Blood Pressure: greater than or equal to (>=) 160mmHg | 0 | 0
  Systolic Blood Pressure: Change from predose greater than (>) 20 mmHg | 11.1 | 0
  Diastolic Blood Pressure: <50 mmHg | 0 | 4.0
  Diastolic Blood Pressure: >=100 mmHg | 0 | 0
  Diastolic Blood Pressure: Change from predose >20 mmHg | 14.8 | 0
  Heart Rate: <40 beats per minute (bpm) | 0 | 0
  Heart Rate: >115 bpm | 0 | 0

4. Primary Outcome: Percentage of Participants With Markedly Abnormal Criteria for 12-lead Safety Electrocardiogram (ECG) Parameters
Time Frame: Study Day 1 up to Study Day 4
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-925 112 mg
Number analyzed (Participants) | 27 | 25
percentage of participants
  PR Interval, Aggregate: <=80 millisecond (msec) | 0 | 0
  PR Interval, Aggregate: >=200 msec | 3.7 | 0
  QRS Duration, Aggregate: <= 80 msec | 11.1 | 12.0
  QRS Duration, Aggregate: >=180 msec | 0 | 0
  QTcF Interval, Aggregate: <=300 msec | 0 | 0
  QTcF Interval, Aggregate: >500 msec | 0 | 0
  QTcF Interval, Aggregate: >=30 change from baseline and >450 msec | 0 | 0
  Heart Rate: <40 bpm | 0 | 0
  Heart Rate: >115 bpm | 0 | 0

5. Secondary Outcome: Ceoi: Observed Plasma Concentration at the End of Infusion for TAK-925
Time Frame: Treatment Periods 1 and 2: Study Day 1 pre-dose, at multiple time points (up to 9 hours) after start of infusion, and at multiple time points (up to 15 hours) after end of infusion
Population: The Pharmacokinetic (PK) analysis set included participants who receive at least 1 dose of study drug and who had at least 1 measurable plasma concentration of TAK-925 (or its metabolites). Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | TAK-925 112 mg
Number analyzed (Participants) | 18
nanogram per milliliter (ng/mL) | 222.0 (31.3)

6. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-925
Time Frame: as for outcome 5
Population: The PK analysis set included participants who receive at least 1 dose of study drug and who had at least 1 measurable plasma concentration of TAK-925 (or its metabolites). Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | TAK-925 112 mg
Number analyzed (Participants) | 18
nanogram*hour per milliliter (ng*h/mL) | 2253 (22.5)

7. Secondary Outcome: AUC Last: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for TAK-925
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | TAK-925 112 mg
Number analyzed (Participants) | 19
ng*h/mL | 2265 (22.3)

ADVERSE EVENTS:
Time Frame: TEAEs were adverse events that started after the start of the first infusion of study treatment (Study Day 1) up to Study Day 11
Description: At each visit the investigator had to document any occurrence of adverse events, including clinically significant abnormal clinical laboratory, vital sign or ECG values. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-925 112 mg
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 2/27 | 5/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | TAK-925 112 mg (N=25)
Headache (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT04091438/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT04091438/SAP_001.pdf